CLINICAL TRIAL: NCT06458465
Title: Clinical Study Evaluating the Impact of Curcumin and Pentoxiphylline on Patients With Chronic Kidney Disease
Brief Title: Impact of Curcumin and Pentoxiphylline on Chronic Kidney Disease Patients
Acronym: CKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Collaborators: Tanta University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0107820
Record Dates: First submitted 2024-05-24; First posted 2024-06-13 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2023-09

CONDITIONS: Chronic Kidney Disease
Keywords: Curcumin; Pentoxiphylline; Chronic Kidney Disease
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Curcumin; Pentoxifylline

STUDY DESIGN:
Intervention Model Description: Open labelled, three-arms, randomized, non-placebo, controlled, parallel clinical trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- No Intervention: Patients receiving no intervention (No Intervention): Group one will not receive add-on therapy; they will receive standard care only.
- Active Comparator: Patients receiving curcumin (Active Comparator): Group two will receive curcumin as an add-on therapy on daily basis
  Interventions: Dietary Supplement: Curcumin
- Active Comparator: Patients receiving pentoxiphylline (Active Comparator): Group three will receive pentoxiphylline as an add-on therapy on daily basis
  Interventions: Drug: Pentoxifylline 400 MG

INTERVENTIONS:
Dietary Supplement: Curcumin — - Curcumin capsules 500 mg twice daily for 6 months
  Arms: Active Comparator: Patients receiving curcumin
Drug: Pentoxifylline 400 MG — - Pentoxifylline 400 mg twice daily for 6 months.
  Other Names: Trental
  Arms: Active Comparator: Patients receiving pentoxiphylline

SUMMARY:
The aim of the study is to evaluate the impact of turmeric and pentoxiphylline on serum levels of protein-bound uremic toxin (p-cresyl sulfate), oxidative stress biomarker level (Malonaldehyde), inflammatory biomarker level (Highly sensitive C-reactive protein). In addition to the evaluation of its effect on metabolic profile and disease progression in chronic kidney disease patients.

DETAILED DESCRIPTION:
1. Ethical committee approval has been obtained from Ethics committee of Faculty of Medicine, Alexandria University.
2. All participants should agree to take part in this clinical study and will provide informed consent.
3. Sixty chronic kidney disease patients will be recruited from the Kidney and Urology Center (KUC) and Alexandria main university hospital (AMUH).

   The 60 participants will be randomly assigned into 3 arms.

   Group 1 (Control group; n=20): Patients will be treated with standard care only for 6 months. Group 2 (n=20): Patients will be treated with the same standard care plus curcumin capsules 500 mg twice daily for 6 months. Group 3 (n=20): Patients will be treated with the same standard care plus pentoxiphylline 400 mg twice daily for 6 months.
4. All patients will be submitted to :

   Full patient history and clinical examination. Blood withdrawal in order to conduct lab work.
5. Patients demographic data will be recorded with respect to age, weight and other co-morbidities.
6. Statistical tests appropriate to the study design will be conducted to evaluate the significance of the results.
7. Results, conclusion, discussion and recommendations will be given.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old.
* Both sexes.
* Non-hemodialysis CKD patients (Stage III -V)
* Patients matched in the duration of CKD.
* Patients with albumin-to-creatinine ratio ≥ 30 mg/g.
* Patients with serum Potassium < 5 mEq/L

Exclusion Criteria:

* Patients with elevated level of potassium ≥ 5 mEq/L.
* Patients with cancer.
* Patients with kidney stones and urinary tract infection.
* Patients with bleeding disorder.
* History of drug allergy to study medications.
* Pregnant and breastfeeding women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-09-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
The change in p-cresyl sulphate biomarker | 6 Months
  the change in biological markers (pCS).
The change in high senstive c-reactive protiem biomarker | 6 Months
  the change in biological marker (hs-CRP)
The change in malonaldehyde biomarker | 6 Months
  the change in biological marker (MDA)
The change in estimated glomerular filtration rate | 6 Months
  the change in eGFR
The change in serum creatinine and BUN | 6 Months
  the change in values of serum creatinine and BUN
The change in proteinuria | 6 Months
  the change in value of proteinuria

SECONDARY OUTCOMES:
Number of participants losing the follow up | 6 Months
  Non-adherence to study medications, loss of follow-up, existence of intolerable side effects, shifting of patients to dialysis, changing of standard care medications and death.

CONTACTS AND LOCATIONS:
Locations (1):
- Nada Mustafa Kamel, Alexandria, Alexandria Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No